CLINICAL TRIAL: NCT06705933
Title: Effect of Kinesiotaping on Postpartum Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Sobhy Kamal mohareb, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005017
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability exercise and myofascial release group (Active Comparator): The participants will receive core stability exercise and myofascial release for 20 min three times per week for 8 weeks.
  Interventions: Other: Core stability exercise; Other: Myofascial release
- Kinesiotaping, in addition to core stability exercise and myofascial release group (Experimental): The participants will receive kinesiotaping, in addition to core stability exercise and myofascial release for 8 weeks
  Interventions: Other: Core stability exercise; Other: Myofascial release; Other: Kinesiotaping

INTERVENTIONS:
Other: Core stability exercise — Lumbo-pelvic stabilizing exercises (posterior pelvic tilt, bilateral hip abduction, bilateral knee raise, bridging, hip shrugging) will be performed three times per week for eight weeks.
Other: Myofascial release — The participants will receive myofascial release technique for 20 min for 3 times per week for 8 weeks.
Other: Kinesiotaping — The participants will receive Kinesio-Taping over the sacroiliac joint and the hip region. Following a test trial of a small patch for 24 hours, they will be instructed to keep the tape on for 48 hours (it will be replaced after 48 hours) . It will be applied for 8 weeks.
  Arms: Kinesiotaping, in addition to core stability exercise and myofascial release group

SUMMARY:
The purpose of this study is to investigate the effect of kinesiotaping on pelvic girdle pain in postpartum women.

DETAILED DESCRIPTION:
Pregnancy-related pain in the SIJ, lumbosacral region, pubic symphysis, or in any combination of these joints has been coined as pelvic girdle pain (PGP) and has been estimated to affect almost half of all pregnant women. Women with PGP have an increased risk of prenatal anxiety, depressive symptoms and postpartum depression compared with healthy pregnant women.

Kinesio Taping is rehabilitative technique used to facilitate the body's natural healing process while providing support and stability to muscles and joints, without restricting their range of motion. Enhanced rehabilitation is thought to be the effect of stimulated reactivation, proprioceptive training, reduced pain, stimulation of correct movement patterns, and reduction of muscle imbalance.

Kinesio Taping (KT) method has been used to decrease and prevent pain in women suffering from pregnancy related low back pain because of increased muscle relaxation while taping is applied. However, there is lack of knowledge regarding the effect of kinesiotaping on PGP in postpartum women.

Therefore, this study will be conducted to provide physiotherapists with a scientific updated knowledge, concerning the effect of kinesiotaping on pain, level of disability and lumbar flexion and extension ROM in pelvic girdle pain in postpartum women, aiming to improve ADLs of postpartum women. This study may expand the role of physiotherapy in women's health

ELIGIBILITY:
Inclusion Criteria:

* All post-partum women < 4 months postnatal having pelvic girdle pain.
* They will be diagnosed using Faber test, and active straight leg raising test.
* Their ages will range from 25 to 35 years.
* Their body mass index (BMI) less than 30 kg/ m².

Exclusion Criteria:

* Pregnant women or planning for pregnancy.
* Cardiovascular diseases.
* Previous spinal surgery.
* History of skeletal deformity.
* Participation at any other exercise training program during this study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | 8 weeks
  Visual analog scale will be used to assess pain level in each woman in both groups before and after the treatment program. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
Measurement of disability level | 8 weeks
  The Oswestry disability index will be used to assess function disability. It is a questionnaire consisting of 10 questions about the impact of low back pain on daily life. Unlike other outcome measures in which a higher score is typically a better score, a higher score on the ODI indicates a greater level of disability, according to the following scoring criteria:0-4: No disability; 5-14: Mild disability; 15-24: Moderate disability; 25-34: Severe disability; 35-50: Completely disabled
Assessment of lumbar flexion range of motion (ROM) | 8 weeks
  Lumbar flexion ROM will be tested by using the inclinometer. The T12 spinous process and the sacral midpoint as landmarks for inclinometer placement. These original landmarks will be modified to the spinal interspaces between T12-L1 and L5-S1 as an attempt to isolate the lumbar spine, and because it was thought that these landmarks are more easily palpated.
  The trial will begin with the patient in a neutral standing position, with the lumbar spine exposed and feet placed shoulder width apart. The subject will be asked to bend forward as far as possible, keeping their legs straight. This point will be entered as a maximum flexion. Normal lumbar flexion (40-60 degrees).
Assessment of lumbar extension range of motion (ROM) | 8 weeks
  Lumbar extension ROM will be tested by using the inclinometer. The T12 spinous process and the sacral midpoint as landmarks for inclinometer placement. These original landmarks will be modified to the spinal interspaces between T12-L1 and L5-S1 as an attempt to isolate the lumbar spine, and because it was thought that these landmarks are more easily palpated.
  The trial will begin with the patient in a neutral standing position, with the lumbar spine exposed and feet placed shoulder width apart. The patient will then be asked to extend back as far as possible with their hands on their hips. This point will be entered as maximal extension. Normal lumbar extension (20-35 degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Elham Hassan, PHD, Study Director — Cairo University; Abeer Eldeeb, Professor, Study Chair — Cairo University
Locations (1):
- Mariam Sobhy kamal, Cairo, Egypt